CLINICAL TRIAL: NCT03674567
Title: Phase 1/2 Dose-Escalation and Expansion Study of FLX475 Alone and in Combination with Pembrolizumab in Advanced Cancer
Brief Title: Dose Escalation and Expansion Study of FLX475 Monotherapy and in Combination with Pembrolizumab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RAPT Therapeutics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FLX475-02; KEYNOTE-877 (Other: Merck Sharp & Dohme LLC); MK-3475-877 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Advanced Cancer
Keywords: Non-small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Breast Cancer; Urothelial Carcinoma; Nasopharyngeal Carcinoma; Cervical Cancer; Lymphoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Carcinoma, Transitional Cell; Nasopharyngeal Carcinoma; Uterine Cervical Neoplasms; Lymphoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1a: Monotherapy Dose Escalation (Experimental): Eligible subjects will be enrolled in sequential cohorts treated with successively higher doses of FLX475 as monotherapy.
  Interventions: Drug: FLX475
- Part 1b: Combination Dose Escalation (Experimental): Eligible subjects will be enrolled in sequential cohorts treated with successively higher doses of FLX475 in combination with pembrolizumab.
  Interventions: Drug: FLX475; Drug: pembrolizumab (KEYTRUDA®)
- Part 2a: Monotherapy Expansion Cohorts (Experimental): Eligible subjects will be initially enrolled in Stage 1 of parallel expansion cohorts of FLX475 as monotherapy; additional subjects in each cohort may be enrolled in Stage 2.
  Interventions: Drug: FLX475
- Part 2b: Combination Expansion Cohorts (Experimental): Eligible subjects will be initially enrolled in Stage 1 of parallel expansion cohorts of FLX475 in combination with pembrolizumab; additional subjects in each cohort may be enrolled in Stage 2.
  Interventions: Drug: FLX475; Drug: pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: FLX475 — tablet
Drug: pembrolizumab (KEYTRUDA®) — IV infusion
  Arms: Part 1b: Combination Dose Escalation; Part 2b: Combination Expansion Cohorts

SUMMARY:
This clinical trial is a Phase 1/2, open-label, sequential-group, dose-escalation and cohort expansion study to determine the safety and preliminary anti-tumor activity of FLX475 as monotherapy and in combination with pembrolizumab.

The study will be conducted in 2 parts, a dose-escalation phase (Part 1) and a cohort expansion phase (Part 2). In Part 1 of the study, subjects will be enrolled in sequential cohorts treated with successively higher doses of FLX475 as monotherapy or in combination with pembrolizumab. In Part 2 of the study, subjects will be initially enrolled in Stage 1 of parallel expansion cohorts of FLX475 as monotherapy or in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Documented advanced or metastatic cancer ineligible for standard therapies with one of the following histologies

  * Dose Escalation: non-small cell lung cancer, head and neck squamous cell carcinoma, nasopharyngeal carcinoma, metastatic triple negative breast cancer, urothelial carcinoma, gastric cancer, esophageal carcinoma, cervical cancer, classical Hodgkin lymphoma
  * Dose Expansion: nasopharyngeal carcinoma, lymphoma, head and neck squamous cell carcinoma, cervical cancer, non-small cell lung cancer, triple-negative breast cancer
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Evaluable disease at baseline (at least one measurable target lesion by imaging for expansion cohorts)
* Tumor available for biopsy

Exclusion Criteria:

* History of allergy or severe hypersensitivity to biologic agents
* History of Grade 3-4 immune-related adverse events leading to discontinuation of prior immuno-oncology treatment
* Active autoimmune disease or serious autoimmune disease within past 2 years requiring systemic therapy
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, (non-infectious) pneumonitis that required steroids, or symptoms of active pneumonitis
* Prior allogeneic hematopoietic stem cell transplant within 5 years, or prior allogeneic organ transplant
* Active graft-versus-host disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of FLX475 as a single agent and in combination with pembrolizumab measured by the incidence of adverse events, including dose-limiting toxicities and maximum tolerated dose | Approximately 18 weeks
Overall response rate in subjects treated with FLX475 as a single agent and in combination with pembrolizumab | Through study completion (approximately 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: William Ho, MD, PhD, Study Director — RAPT Therapeutics, Inc.
Locations (35):
- United States (19):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - University of California, Los Angeles JCCC Clinical Research Unit, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Comprehensive Hematology and Oncology, LLC, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Louisville Hospital/James Graham Brown Cancer Center, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Quantum Santa Fe, Santa Fe, New Mexico
  - New York Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington
- Australia (2):
  - Austin Hospital, Heidelberg, Victoria
  - Linear Clinical Research Limited, Nedlands, Western Australia
- Hong Kong (3):
  - Queen Mary Hospital - Lymphoma, High West
  - Queen Mary Hospital, High West
  - Prince of Wales Hospital, Shatin
- South Korea (5):
  - Chungbuk National University Hospital, Jungbuk
  - Seoul National University, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Meidcal Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (2):
  - King Chulaongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No